CLINICAL TRIAL: NCT06441058
Title: Influence of the Timing of Post-endodontic Restoration Placement on the Survival of Root Canal-treated Teeth
Brief Title: Retrospective Database Study: Influence of Post-endodontic Restoration Placement on Survival of Root Canal-treated Teeth
Status: Completed | Type: Observational
Sponsor: University of Göttingen (Other)
Responsible Party: Principal Investigator, Philipp Kanzow, Prof. Dr. med. dent., Dr. rer. medic., Senior Lecturer, University Medical Center Goettingen
Other Study IDs: Timing-post-endodontic; 20/2/20 (Other: Local Ethics Commission)
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Root Canal Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Indirect post-endodontic restorations: Indirect post-endodontic restorations (e.g. crown, partial crown).
  Interventions: Other: No patient treatment is associated with the study

INTERVENTIONS:
Other: No patient treatment is associated with the study — No patient treatment is associated with the study.

SUMMARY:
The aim of this study is to assess the influence (i.e. type and timing) of post-endodontic restorations on the survival of root canal-treated teeth and to determine the influence of patient-, tooth-, treatment-, and restoration-specific parameters on longevity.

Patients who received a root-canal treatment between 1998 and 1999 with subsequent placement of an indirect restoration (e.g. crown, partial crown) will be retrospectively analyzed. Patient-, tooth-, treatment-, and restoration-specific parameters will be obtained from digital and paper-based dental records.

Survival and success of the root-canal treatments will be assessed using Kaplan-Meier statistics. Mean annual failure rates (mAFR) and median survival time will be calculated (Kaplan-Meier statistics). Potential predictive factors will be tested using log-rank tests and multi-variate Cox-regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received a root-canal treatment followed by the placement of an indirect post-endodontic restoration (e.g. partial crowns, crowns) within the Department of Preventive Dentistry, Periodontology and Cariology between 1998 and 1999.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received a root-canal treatment followed by the placement of an indirect post-endodontic restoration (e.g. partial crowns, crowns) within the Department of Preventive Dentistry, Periodontology and Cariology between 1998 and 1999.
Sampling Method: Non-Probability Sample
Enrollment: 541 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Success of endodontic treatment | 1998-2023
  Success is defined as the time-interval without a subsequent endodontic re-intervention or extraction of the tooth.

SECONDARY OUTCOMES:
Survival of the tooth | 1998-2023
  Survival of the tooth is defined as the time-interval without extraction of the tooth.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Göttingen, Dept. of Preventive Dentistry, Periodontology and Cariology, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No